CLINICAL TRIAL: NCT02245646
Title: Subjektiv Verzerrter Höreindruck Nach Stapedotomie
Brief Title: Distortion Product After Stapedotomy Surgery
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AH-RG_03_06_2014
Record Dates: First submitted 2014-09-10; First posted 2014-09-19 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Distorted Sound Perception

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control group: No indication for stapedotomy
- Distortion positive: Subjects after stapedotomy perceiving sound distortions
- Distortion negative: Subjects after stapedotomy not perceiving sound distortions.

SUMMARY:
This study aims at capturing for the first time at which frequencies and sound intensities hearing distortions are perceived after successful stapedotomy surgery. Also, the portion of patients perceiving these sound distortions and the length of time over which the distortions occur are assessed.

DETAILED DESCRIPTION:
If the stapes footplate is fixed in position, e.g. by otosclerosis, rather than being normally mobile, a conductive hearing loss results. This conductive hearing loss is usually compensated with hearing aids or through stapedotomy. During stapedotomy, the diseased stapes bone is removed and is replaced with a piston prosthesis that conveys the sound stimulus from the incus to the footplate of the removed stapes.

After surgery subjects sometimes state that the quality of sound is suboptimal, even though their hearing ability has improved significantly. Some subjects subjectively hear distorted sounds, which often disappear several weeks after surgery.

This study aims at capturing for the first time at which frequencies and sound intensities these distortions are perceived. Additionally, the portion of patients perceiving these sound distortions and the length of time over which the distortions occur are assessed.

ELIGIBILITY:
Inclusion Criteria:

* indication for stapedotomy
* written consent given

Exclusion Criteria:

* not mentally able to give written consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Control group: Healthy volunteers are recruited by flyers that are displayed in the waiting zones of the ENT clinic.
  Subjects with stapedotomy: Patients are being asked by the examining MD as soon as the indication for stapedotomy is proven.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
Change of distorted sound perception after stapedotomy surgery | 7 to 14 days post surgery; 21 to 25 days post surgery; 3, 6 and 12 months post surgery
  A psychoacoustic audiometric tests is performed; subjects are asked to press a button if the sound they hear is distorted, and this is tested at different frequencies and different level of loudness.

SECONDARY OUTCOMES:
Questionnaire on quality of hearing after Stapedotomy (APOSE) | 7 to 14 days post surgery; 21 to 25 days post surgery; 3, 6 and 12 months post surgery
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Huber, Prof., Study Chair — USZ
Locations (1):
- Zurich University Hospital, Division of Otorhinolaryngology, Head and Neck Surgery, Zurich, Switzerland